CLINICAL TRIAL: NCT05198180
Title: Comparative Study Between Topical30%Potassium Hydroxide Solution and Topical 45% Hydrogen Peroxide Solution in Treatment of Plantar Warts
Brief Title: Treatment of Plantar Warts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samar Sayed Ahmed, Principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sohag-Mes-21-11-07
Record Dates: First submitted 2021-12-26; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Plantar Wart

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium hydroxide group (Active Comparator): Patients with plantar warts will apply topical 30% potassium hydroxide solutions on warts
  Interventions: Drug: Topical 30%Potassium hydroxide solution
- Hydrogen peroxide group (Active Comparator): Patients with plantar warts will use topical 45% hydrogen peroxide solution on warts
  Interventions: Drug: Topical 45% hydrogen peroxide solution

INTERVENTIONS:
Drug: Topical 30%Potassium hydroxide solution — Patients will apply the solution every day under occlusion for 3 months
  Arms: Potassium hydroxide group
Drug: Topical 45% hydrogen peroxide solution — Patients will apply the solution every day under occlusion
  Arms: Hydrogen peroxide group

SUMMARY:
This study is to compare the efficacy and safety of topical 30% potassium hydroxide solution and topical 45% hydrogen peroxide solution in treatment of plantar warts.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis by clinical and dermoscopic examination of plantar warts

Exclusion Criteria:

* history of hypersensitivity to any component used in this study
* pregnancy and breastfeeding
* patients who receive immune suppressive therapy
* patients who received any wart treatments during the last 2 months before enrollent in the study
* patients who refused participation in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the size of the plantar warts | 12 weeks after end of treatment
  Decrease in the size of warts measured by a ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No